CLINICAL TRIAL: NCT04403178
Title: Prediction of Hip Displacement in Children With Cerebral Palsy Among Patients Participating in the Danish Cerebral Palsy Follow-up Program
Brief Title: Prevention of Hip Displacement in Children With Cerebral Palsy in Denmark
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mette Røn Kristensen (Other)
Responsible Party: Sponsor-Investigator, Mette Røn Kristensen, Regional coordinator for CPOP in the capital region of Denmark, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: P-2019-143 2
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Child; Cerebral Palsy; Radiography; Hip Dislocation; Hip Displacement; Prospective Studies
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children who develops hip displacement: Patient group 1 includes children who developed a Migration Percentage of > 40 % in either hip over a follow-up period of three years.
- Children who do not develops hip displacement: Patient group 2 includes children who did not develop a Migration Percentage of > 40 % on either hip over a follow-up period of three years
  Interventions: Diagnostic Test: Radiographic examination with a Migration of > 40 %

INTERVENTIONS:
Diagnostic Test: Radiographic examination with a Migration of > 40 % — Radiographic examination
  Groups: Children who do not develops hip displacement

SUMMARY:
Children with cerebral palsy have an increased risk of hip dislocation, which is a painful and severe complication of cerebral palsy. The 20-years evaluation of the Swedish surveillance programme shows that hip dislocation in children with cerebral palsy can be prevented with regular clinical and radiographic examination and early intervention.

We would like to determine the individual risk for hip displacement for Danish children with CP in The Danish Cerebral Palsy Follow-up Program. This could be a valuable clinical tool in deciding on further follow-up and treatment.

DETAILED DESCRIPTION:
Migration percentage (MP) which is measured from the pelvis radiograph is commonly used to assess lateral displacement of the femoral head and is being used in the Swedish and in the Danish surveillance programme. Most children with an MP > 40 % need surgery to prevent further displacement and prevent dislocation of the hip. In the Swedish surveillance programme they have developed the Cerebral Palsy Follow-Up Programme (CPUP) hip score as a risk score to determine which children are at high or low risk for hip displacement (MP > 40 %) within five years after first radiographic examination.

The aim of this study is to predict the likelihood that a child with cerebral palsy will develop hip displacement (MI> 40) within three years. The design is a prediction study.

Data will be obtained from the national clinical quality database the Danish Cerebral Palsy Follow-up Program and the Danish National Patient Register.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Gross Motor Function Classification System III to V
* Migration Percentage < 40 % for both hips at the first pelvic radiographic examination

Exclusion Criteria:

* Previous femoral osteotomy
* Previous pelvic osteotomy
* Previous selective dorsal rhizotomy
* Intrathecal baclofen pump treatment
* Children whose diagnosis was not confirmed
* Children who were no longer followed in the children's ward at the hospital
* Children who moved out of the area
* Children who died during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with cerebral palsy in Denmark. Data will be obtained from the national clinical quality database the Danish Cerebral Palsy Follow-up Program and the Danish National Patient Register.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-12-27 (Estimated)

PRIMARY OUTCOMES:
Development of hip displacement or not measured by the Migration Percentage | Follow-up period of three years.
  Migration Percentage (MP) is measured from a pelvis radiograph and is used to assess lateral displacement of the femoral head. A MP < 40 % on either hip is a good outcome, whereas a MP > 40 % on either hip is a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Røn Kristensen, PT, MSc, Principal Investigator — Afsnit 234- 236, Fysio- og ergoterapien, Hvidovre Hospital
Locations (1):
- Fysio- og Ergoterapien, afsnit 234-236, Hvidovre hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermanson M, Hagglund G, Riad J, Rodby-Bousquet E, Wagner P. Prediction of hip displacement in children with cerebral palsy: development of the CPUP hip score. Bone Joint J. 2015 Oct;97-B(10):1441-4. doi: 10.1302/0301-620X.97B10.35978. PMID 26430023
- [Background] Rasmussen HM, Nordbye-Nielsen K, Moller-Madsen B, Johansen M, Ellitsgaard N, Pedersen CR, Rackauskaite G, Engberg H, Pedersen NW. The Danish Cerebral Palsy Follow-up Program. Clin Epidemiol. 2016 Oct 25;8:457-460. doi: 10.2147/CLEP.S99474. eCollection 2016. PMID 27822084
- [Background] Hagglund G, Alriksson-Schmidt A, Lauge-Pedersen H, Rodby-Bousquet E, Wagner P, Westbom L. Prevention of dislocation of the hip in children with cerebral palsy: 20-year results of a population-based prevention programme. Bone Joint J. 2014 Nov;96-B(11):1546-52. doi: 10.1302/0301-620X.96B11.34385. PMID 25371472